CLINICAL TRIAL: NCT00641914
Title: Inhaled Steroid Treatment As Regular Therapy in Early Asthma. A Study on the Effect of Early Intervention With Long-Term Inhaled Budesonide (Pulmicort Turbuhaler ® ) in Newly Diagnosed Asthma.
Brief Title: Inhaled Steroid Treatment as Regular Therapy in Early Asthma
Acronym: START
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Lars-Göran Carlsson, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SD-004-0111; D5254C00111
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Asthma
Keywords: Asthma; Pulmicort; budesonide
MeSH Terms: conditions — Asthma | interventions — Budesonide

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: budesonide
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: budesonide
  Other Names: Pulmicort
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
A study of the effect of the early treatment with Pulmicort of newly diagnosed asthma. Patients will receive either Pulmicort or a non-active treatment for three years. Neither patients or investigators will be aware of the treatment received. After three years of treatment all patients will receive Pulmicort for 2 further years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 6 and 60 years
* diagnosed with asthma within 2 years of starting the study
* Ability to use a Turbuhaler

Exclusion Criteria:

* Symptoms indicating asthma (e.g. wheezing) for more than two years prior to starting the study
* A history of the use of treatments like Pulmicort for more than 30 days per year in the two years before starting the study
* Regular daily treatment for asthma for more than two years before starting the study

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6800 (Estimated)
Dates: Start 1996-10; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Severe asthma related events (SARE) (part A); post-bronchodilator FEV1 % of predicted normal (part B) | At week 6 and12, and every 3 months thereafter

SECONDARY OUTCOMES:
Pre-bronchodilator FEV1 % of predicted normal | At week 6 and12, and every 3 months thereafter
HE: Asthma related events and health care utilisation, and symptom free days (SFD) | At week 6 and12, and every 3 months thereafter
Post-bronchodilator FVC % of predicted | At week 6 and12, and every 3 months thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Romain Pauwels, Study Chair — Steering Committee Chairman; William Busse, Study Chair — Steering Committee Chairman

REFERENCES:
- [Derived] O'Byrne PM, Pedersen S, Lamm CJ, Tan WC, Busse WW; START Investigators Group. Severe exacerbations and decline in lung function in asthma. Am J Respir Crit Care Med. 2009 Jan 1;179(1):19-24. doi: 10.1164/rccm.200807-1126OC. Epub 2008 Oct 31. PMID 18990678